CLINICAL TRIAL: NCT01425879
Title: A Multi-Institutional Phase II Study of the Akt Inhibitor MK-2206 in Refractory Biliary Cancers
Brief Title: MK2206 in Treating Patients With Advanced Refractory Biliary Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02974; NCI-2011-02974 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-10104; OSU 10104; CDR0000698451; OSU 10104 (Other: Ohio State University Comprehensive Cancer Center); 8735 (Other: CTEP); N01CM00070 (NIH); P30CA016058 (NIH)
Record Dates: First submitted 2011-08-27; First posted 2011-08-30 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Advanced Adult Hepatocellular Carcinoma; Localized Non-Resectable Adult Liver Carcinoma; Recurrent Adult Liver Carcinoma; Recurrent Gallbladder Carcinoma; Stage IV Distal Bile Duct Cancer; Stage IV Gallbladder Cancer; Unresectable Extrahepatic Bile Duct Carcinoma; Unresectable Gallbladder Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Gallbladder Neoplasms | interventions — MK 2206

ARMS (1):
- Treatment (Akt inhibitor MK2206) (Experimental): Patients receive Akt inhibitor MK2206 PO on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Other: Diagnostic Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial is studying how well MD2206 works in treating patients with advanced refractory biliary cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the objective response rate (complete and partial response), as defined by the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria, in patients with advanced refractory biliary cancers (BC) receiving Akt inhibitor MK2206 (MK2206).

SECONDARY OBJECTIVES:

I. To determine the frequency and severity of adverse events and tolerability of the regimen in patients with advanced refractory BC receiving MK2206.

II. To determine the overall and progression-free survival of patients with advanced refractory BC receiving MK2206.

III. To determine the presence of genetic mutations of PI3-kinase/ Akt pathway signaling-pathway genes relevant to BC and how these correlate with objective response to treatment with MK2206.

IV. To determine the pharmacokinetic and pharmacogenetic profile as a way of assessing inter-individual variability as well as how these relate to clinical outcomes.

V. To determine genetic variants and mutations in genes encoding drug-metabolizing enzymes and transporters, and genes involved in tumor biology, and how these may be related to response to treatment.

OUTLINE: This is a multicenter study.

Patients receive Akt inhibitor MK2206 orally (PO) on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and periodically during study for pharmacokinetic, pharmacogenetic, and other correlative studies. Previously collected tumor tissue is also analyzed.

After completion of study therapy, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed biliary tract carcinoma that is surgically unresectable

  * Cytological confirmation is not allowed on this study, as tissue is needed for correlative science analysis
  * Either fresh-frozen tissue (FFT) or paraffin-embedded tissue blocks (PETB) will be required from patients before enrolling on this study
  * No biopsies will be required unless there is insufficient tissue or if the PETB available is more than 12 months old
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with spiral CT scan (CT scan slice thickness no greater than 5 mm)

  * Malignant lymph nodes will be considered measurable if they are ≥ 15 mm in short axis
* Patients must have received one prior therapy for metastatic disease

  * No prior Akt inhibitors allowed
* Patients with known brain metastases should be excluded from this clinical trial
* Life expectancy greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =<2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelet count >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT] =< 2.5 x IULN
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (measured or calculated using the Cockroft-Gualt formula)
* Women of childbearing potential and men must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Not pregnant or nursing
* Able to swallow oral tablets
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to Akt Inhibitor MK2206 (MK2206) or other agents used in the study
* Patients with diabetes or in risk for hyperglycemia should not be excluded from trials with MK2206, but the hyperglycemia should be well controlled on oral agents before the patient enters the trial
* Cardiovascular: baseline QTcF > 450 msec (male) or QTcF > 470 msec (female) will exclude patients from entry on study
* Patients with clinically significant bundle branch block or pre-existing clinically significant bradycardia will be excluded from the study
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; or psychiatric illness/social situations that would limit compliance with study requirements
* No concurrent grapefruit or grapefruit juice
* For patients having prior cryotherapy, radiofrequency ablation, ethanol injection, transarterial chemoembolization (TACE), or photodynamic therapy, the following criteria must be met:

  * 6 weeks has elapsed since that therapy
  * Indicator lesion(s) is/are outside the area of prior treatment or, if the only indicator lesion is inside the prior treatment area, there must be clear evidence of disease progression associated with that lesion
  * Edges of the indicator lesion are clearly distinct on CT scanning
  * Prior radiation therapy with or without the use of a fluoropyrimidine as a radiosensitizer in the adjuvant setting will be allowed on study if > 12 weeks have elapsed since therapy
  * Prior palliative radiation therapy will allowed as long as > 4 weeks have elapsed since therapy
* No patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients receiving any medications or substances that are inhibitors or inducers of CYP 450 3A4 are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-04; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanios Bekaii-Saab, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (8):
- United States (8):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Seidman Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between September 2012 and December 2013
Period: Overall Study
Arm/Group | Treatment (Akt Inhibitor MK2206)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 58 [40 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: patients]
  United States | 8
Disease site [Number; unit: patients]
  Intrahepatic | 6
  Gallbladder | 0
  Extrahepatic | 2
ECOG Performance Status [Number; unit: patients] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
  PS 0 defined as Normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  PS 1 defined as Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g. light housework, office work).
  patients
    PS 0 | 2
    PS 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete and Partial Response) as Defined by RECIST 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 4 weeks after completion of study treatment, for total treatment time of up to 1 year
Measure: Number; unit: patients
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 8
patients | 0

2. Secondary Outcome: Frequency of Adverse Events Related to MK-2206
Description: Severity of adverse events is graded according to the NCI CTCAE 4.0.
Time Frame: Up to 4 weeks after completion of study treatment, for total treatment time of up to 1 year
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 8
percentage of patients
  lymphopenia | 75
  rash | 63
  fatigue | 50
  fever | 50
  vomiting | 50
  diarrhea | 50

3. Secondary Outcome: Overall Survival
Description: Analyzed using Kaplan-Meier method.
Time Frame: From study initiation to time of death, assessed up to 4 weeks after completion of study treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 8
months | 3.5 [2.2 to 6.7]

4. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From start of treatment to time of documented progression or death whichever occurs first, assessed up to 4 weeks after completion of study treatment
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 8
months | 1.7 [0.5 to 5.6]

ADVERSE EVENTS:
Time Frame: All patients were evaluable for toxicity from the time of their first treatment with MK2206
Description: NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4 was utilized for Adverse Event reporting.
Arm/Group | Treatment (Akt Inhibitor MK2206)
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=8)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dry Mouth (Gastrointestinal disorders) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3)
Fatigue (General disorders) | 4 (4)
Fever (Blood and lymphatic system disorders) | 4 (4)
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Leukopenia (Investigations) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 6 (6)
Macular Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Mucositis (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less